CLINICAL TRIAL: NCT02447393
Title: A Single Blind, Randomized, Single Oral Dose Study to Compare the Oral Disposition of Levocetirizine When Given Alone (5mg) or as the Racemate (Cetirizine 10mg), and to Investigate the Safety and Tolerability and the Pharmacokinetics of Levocetirizine and Cetirizine, Following a Single Dose in Healthy Japanese Male Subjects
Brief Title: Phase 1 Study of Levocetirizine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 111580
Record Dates: First submitted 2011-06-23; First posted 2015-05-18 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — levocetirizine; Cetirizine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- levocetirizine (Other): Study Drug
  Interventions: Drug: levocetirizine
- cetirizine (Other): Study Drug
  Interventions: Drug: cetirizine
- placebo (Other): Study Drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levocetirizine — levocetirizine
  Arms: levocetirizine
Drug: cetirizine — cetiridine
  Arms: cetirizine
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This is a single center, single blind, single dose, randomized, partial cross-over study to confirm bioequivalence between levocetirizine and cetirizine.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy male subjects aged between 20 and 64 years of age inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies, and other tests.
2. Body weight ≥ 50 kg and BMI within the range 18.50-25.00 kg/m2 inclusive.
3. Non-smokers (at least 6 months).
4. Clinical laboratory tests data obtained at screening meet the following:

   AST(GOT), ALT(GPT), total-bilirubin, BUN, creatinine, uric acid,: below the upper normal range
5. Normal 12-lead EGC finding at screening; QTc interval <450msec
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
2. The subject has an allergy for any drug or idiosyncrasy.
3. The subject has a history of allergic rhinitis.
4. The subject has a history or presence of clinically significant gastrointestinal, hepatic or renal disease or other condition known to interfere with absorption, distribution, metabolism or elimination of drugs.
5. The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
6. The subject has participated in a clinical study with an investigational or a non-investigational drug or device during the previous 4 months.
7. The subject has a history or current conditions of drug abuse or alcoholism.
8. History of regular alcohol consumption exceeding on average, 14 drinks/week (1 drink = 150mL of wine or 360mL of beer or 45mL of 80 proof distilled spirits).
9. The subject is positive for urine drug screening.
10. The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
11. The subject has donated a unit of blood ">400mL" within the previous 4 months or ">200mL" within the previous 1 month.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

PRIMARY OUTCOMES:
AUC0-48 of levocetirizine | predose,0.25,0.5,1,1.5,2,3,4,6,9,12,16,24,36, 48 hours post-dose
  Area Under the time-concentlation curve
Cmax of levocetirizine | predose,0.25,0.5,1,1.5,2,3,4,6,9,12,16,24,36, 48 hours post-dose
  maximum concentration

SECONDARY OUTCOMES:
Number of Adverse events | predose,1,24 48 hours post-dose
Changes in clinical laboratory tests | predose,24,48 hours post-dose
Changes in vital signs | predose,1,24,48 hours post-dose
Changes in 12-lead ECG. | predose,1,24,48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Kagoshima, Japan

REFERENCES:
- [Background] Hiroko Ino, Shigeru Nohda, Shuji Miki, Kastutoshi Hara, Toshiyasu Hirama. Comparison of levocetirizine pharmacokinetics, following a single dose of levocetirizine alone or as cetirizine in Japanese healthy male volunteers . [Jpn J Clin Pharmacol Therapeut]. 2010;41(6):309.
- See also: Results for study 111580 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111580?search=study&study_ids=111580#rs